CLINICAL TRIAL: NCT06404606
Title: Effects of Black Cumin and Turmeric Along With Quantum Acoustic Waves on Inflammatory Markers and Pain in Osteoarthritis.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Society for Rehabilitation of Differently Abled Hospital (Other)
Collaborators: Innovative Health Concepts and Research Center, Lahore,Pakistan (Unknown); Department of Life Sciences, Univeristy of Management and Technology, Lahore.Pakistan. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IHC&RC-DAH
Record Dates: First submitted 2024-05-05; First posted 2024-05-08 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Quantum Acoustic Waves; Black Cumin &Turmeric.
MeSH Terms: conditions — Osteoarthritis | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Black Cumin & Turmeric) (Active Comparator): Participants will receive one capsule of black cumin and turmeric thrice per week (Alternate days) for 12 weeks.
  Interventions: Combination Product: Black cumin and turmeric with Quantum Acoustic Waves (QAW)
- Group B (Black Cumin & Turmeric along with Quantum Acoustic Waves) (Active Comparator): Participants will receive one capsule of black cumin and turmeric along with Quantum Acoustic Waves (QAW) three days per week for 12 weeks
  Interventions: Combination Product: Black cumin and turmeric with Quantum Acoustic Waves (QAW)
- Group C (Quantum Acoustic Waves) (Active Comparator): Participants will receive Quantum Acoustic Waves (QAW) three days per week for 12 weeks
  Interventions: Combination Product: Black cumin and turmeric with Quantum Acoustic Waves (QAW)

INTERVENTIONS:
Combination Product: Black cumin and turmeric with Quantum Acoustic Waves (QAW) — Black cumin and turmeric are known to be helpful in reduction of inflammation of human body so it will be used in combination with Quantum Acoustic Waves (QAW) to determine effects on initial degenerative changes in osteoarthritis.

SUMMARY:
Osteoarthritis is a chronic inflammatory disease that directly affects the quality of life and financial burden. The understanding of the mechanism and available intervention strategies can not minimize its incidence that increased by 1/10 since 1990. The combination of black cumin and turmeric with sound waves is not well known.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is characterized by insult of the joint involving structural and functional modifications including cartilage rupture, bone deterioration and spur formation; presented with pain, inflammation, joint functional limitation. It is estimated that incidence of osteoarthritis is around 20%. Indeed, it is estimated that incidence is higher in Asia and middle east countries (16-29%) as compared to Europe (10-17%) and north America (12-21%). The aggravating symptoms progress and ultimately cause disability, decline quality of life and put economic burden. Various factors involve in the pathophysiology of OA such as mechanical, inflammatory, metabolic, ageing and genetics that causing structural change and functional limitation along with chronic pain. Nevertheless, there are advancement happening about understanding of the basic mechanism of OA. However, low grade inflammation of the synovial lining is currently considered a major contributing factor that play essential role in understanding the pathophysiology; Moreover, adaptive central immunological mechanism is recognized pivotal in tissue inflammation and destruction. The low-grade inflammation and sensitivity of central nervous system progress to be the factor of chronic pain in OA. In particular, the definition of OA now needs to be renewed and considered as multifactor joint disorder that mainly occurs due to metabolic and inflammatory alteration that causes damage of the joints. Therefore, therapeutic interventions suggested for the management of OA are directly influenced by the current understating of OA pathophysiology. So, various inflammatory cytokines increased in OA tissues such as interleukin (IL)-1, IL,6, IL-15, IL-17, IL-18, and Tissue necrotic factor (TNF). It has been proven that black cumin contributes to human body by its anti-inflammatory and anti-nociceptive properties. Moreover, sound waves can stimulate fluid to mobilize through the body and brain and bring oxygen and essential nutrients to the tissue. Similarly, A low-intensity pulsed ultrasound that uses sound waves is considered effective in reduction of inflammation.

As per the researcher's knowledge, there is limited literature available to determine the effect of turmeric and black cumin on inflammation but, there is very little known about the quantum acoustic waves on inflammation, so this study aims to determine the effects of quantum acoustic waves with black cumin and turmeric.

ELIGIBILITY:
Inclusion Criteria:

* Both genders age between 45 to 60 years.
* Rheumatoid Arthritis (RA) negative.
* C-reactive protein (CRP)negative.
* Erythrocyte Sedimentation Rate (ESR) below 30.
* No intake of Anti-inflammatory drugs (NSAIDS, steroids) during the last 02 weeks.
* Grade 2 and Grade 3 Osteoarthritis as per kellegran criteria.
* Body Mass Index (BMI) between 18.5 kg/m2 to 29.9 kg/m2.
* Vitamin D above 30 ng/dl.

Exclusion Criteria:

* Infective arthritis.
* Reactive arthritis.
* Major Gastrointestinal or cardiovascular disease/disorder.
* Musculoskeletal injury or disorder that limits participation.
* Patients who are not willing to participate.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Inflammatory Markers | Baseline (0-week) and 12th week
  The blood sample will be taken for assessment of Inflammatory cytokines interleukin (IL)-6, IL,10, IL-17, Tissue necrotic factor (TNF), Complete Blood Count (CBC), CRP, ESR, RA factor, Anti-CCP and Vitamin D for functional parameters.

SECONDARY OUTCOMES:
Pain | Baseline (0-week), 4-week, 8-week & 12-week.
  The Standardized Numeric Pain rating Scale (NPRS) will be used for pain assessment of participants. The patients will instruct to rate its pain from 0 to 10. The score interpreted as no pain (0-level) to highest pain (10) where it is further categorized as mild (1-3), moderate (4-7) and severe (8-10).
Knee Injury and Osteoarthritis Outcome Score | Baseline (0-week), 4-week, 8-week & 12-week.
  KOOS questionnaire is self-administered questionnaire that will be used to assess five domains of the participants include pain, symptoms, activities of daily livings, sports and recreational function and knee related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Faheem Afzal, *PhD, Principal Investigator — PSRD Hospital/IHC&RC
Locations (1):
- Innovative Health Concepts & Research Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] March L, Cross M, Lo C, Arden NK, Gates L, Leyland K, et al. Osteoarthritis: A Serious Disease: Submitted to the US Food and Drug Administration. 2016.
- [Result] Safiri S, Kolahi AA, Smith E, Hill C, Bettampadi D, Mansournia MA, Hoy D, Ashrafi-Asgarabad A, Sepidarkish M, Almasi-Hashiani A, Collins G, Kaufman J, Qorbani M, Moradi-Lakeh M, Woolf AD, Guillemin F, March L, Cross M. Global, regional and national burden of osteoarthritis 1990-2017: a systematic analysis of the Global Burden of Disease Study 2017. Ann Rheum Dis. 2020 Jun;79(6):819-828. doi: 10.1136/annrheumdis-2019-216515. Epub 2020 May 12. PMID 32398285
- [Result] Cui A, Li H, Wang D, Zhong J, Chen Y, Lu H. Global, regional prevalence, incidence and risk factors of knee osteoarthritis in population-based studies. EClinicalMedicine. 2020 Nov 26;29-30:100587. doi: 10.1016/j.eclinm.2020.100587. eCollection 2020 Dec. PMID 34505846
- [Result] Abramoff B, Caldera FE. Osteoarthritis: Pathology, Diagnosis, and Treatment Options. Med Clin North Am. 2020 Mar;104(2):293-311. doi: 10.1016/j.mcna.2019.10.007. Epub 2019 Dec 18. PMID 32035570
- [Result] Hu Y, Chen X, Wang S, Jing Y, Su J. Subchondral bone microenvironment in osteoarthritis and pain. Bone Res. 2021 Mar 17;9(1):20. doi: 10.1038/s41413-021-00147-z. PMID 33731688
- [Result] van den Bosch MHJ. Osteoarthritis year in review 2020: biology. Osteoarthritis Cartilage. 2021 Feb;29(2):143-150. doi: 10.1016/j.joca.2020.10.006. Epub 2020 Nov 24. PMID 33242602
- [Result] Geyer M, Schonfeld C. Novel Insights into the Pathogenesis of Osteoarthritis. Curr Rheumatol Rev. 2018;14(2):98-107. doi: 10.2174/1573397113666170807122312. PMID 28782470
- [Result] Kulkarni P, Martson A, Vidya R, Chitnavis S, Harsulkar A. Pathophysiological landscape of osteoarthritis. Adv Clin Chem. 2021;100:37-90. doi: 10.1016/bs.acc.2020.04.002. Epub 2020 May 29. PMID 33453867
- [Result] Geraghty T, Winter DR, Miller RJ, Miller RE, Malfait AM. Neuroimmune interactions and osteoarthritis pain: focus on macrophages. Pain Rep. 2021 Mar 9;6(1):e892. doi: 10.1097/PR9.0000000000000892. eCollection 2021. PMID 33981927
- [Result] Jang S, Lee K, Ju JH. Recent Updates of Diagnosis, Pathophysiology, and Treatment on Osteoarthritis of the Knee. Int J Mol Sci. 2021 Mar 5;22(5):2619. doi: 10.3390/ijms22052619. PMID 33807695
- [Result] Coaccioli S, Sarzi-Puttini P, Zis P, Rinonapoli G, Varrassi G. Osteoarthritis: New Insight on Its Pathophysiology. J Clin Med. 2022 Oct 12;11(20):6013. doi: 10.3390/jcm11206013. PMID 36294334
- [Result] Amin B, Hosseinzadeh H. Black Cumin (Nigella sativa) and Its Active Constituent, Thymoquinone: An Overview on the Analgesic and Anti-inflammatory Effects. Planta Med. 2016 Jan;82(1-2):8-16. doi: 10.1055/s-0035-1557838. Epub 2015 Sep 14. PMID 26366755
- [Result] Altman J. Information processing concerning moving sound sources in the auditory centers and its utilization by brain integrative and motor structures. Auditory pathway: structure and function. 1988:349-54.
- [Result] Xu M, Wang L, Wu S, Dong Y, Chen X, Wang S, Li X, Zou C. Review on experimental study and clinical application of low-intensity pulsed ultrasound in inflammation. Quant Imaging Med Surg. 2021 Jan;11(1):443-462. doi: 10.21037/qims-20-680. PMID 33392043